CLINICAL TRIAL: NCT00386464
Title: Noninvasive Ventilation in ALS Patients With Mild Respiratory Involvement
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HL 67887-03
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2007-11-09 (Estimated); Status verified 2007-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: bipap; lou gehrigs disease; motor neuron disease; respiratory muscles
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: noninvasive positive pressure ventilation

SUMMARY:
Non-invasive ventilation or BiPAP®, which is a form of breathing support delivered through a facemask, is a successful treatment for the respiratory complications of amyotrophic lateral sclerosis (ALS). It has been shown to prolong survival, improve quality of life, and improve cognitive function. It is widely used among patients with ALS who have advanced breathing difficulties. It is not known whether there is benefit to using non-invasive ventilation earlier in the disease course.

There is evidence that non-invasive ventilation may slow down the decline in breathing function. If this were true then it would make sense to start non-invasive ventilation use earlier than the current clinically accepted practices.

The purpose of this study is to determine whether using non-invasive ventilation early in the course of disease can slow the decline in breathing function.

Patients remain in the study for 6 months and are asked to make 7 clinic visits during which time they will undergo pulmonary function tests and complete questionnaires.

DETAILED DESCRIPTION:
This is a randomized, crossover trial for patient with ALS and mild respiratory involvement. Patients with forced vital capacity above 60% of the predicted value can join. Patients will be assigned to either start using non-invasive ventilation at night or continue their usual care. After three months, patients will switch over to the other treatment group. For example, a patient who was initially assigned to continue their usual care would begin using non-invasive ventilation after three months.

ELIGIBILITY:
Inclusion Criteria:

* Probable or definite ALS by El Escorial criteria
* age >17 years
* FVC >60
* minimal respiratory symptoms (no orthopnea or dyspnea at rest)
* ability to provide informed consent

Exclusion Criteria:

* Presence of another neurodegenerative disease
* arterial CO2 above 45 mmHg
* O2 below 60 mmHg
* coexisting chronic lung disease unrelated to ALS
* presence of an unstable medical condition such as coronary artery disease, liver failure, renal failure or cancer in the 30 days preceding enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2002-04; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Decline in forced vital capacity

SECONDARY OUTCOMES:
quality of life
respiratory quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Noah Lechtzin, MD, Principal Investigator — Johns Hopkins University; Charles M Wiener, MD, Study Chair — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- See also: Johns Hopkins ALS Center — http://www.hopkinsneuro.org/ALS/clinical_trials.cfm